CLINICAL TRIAL: NCT03480893
Title: Cost-effectiveness of Small Size Interarcuair Decompression Versus Extended Decompression in Patients With Intermittent Neurogenic Claudication (Size-study): a Multi-center, Double-blinded Randomized Controlled Trial
Brief Title: Cost-effectiveness of Small Size Interarcuair Decompression Versus Extended Decompression in Patients With Intermittent Neurogenic Claudication
Acronym: Size
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Park MC (Unknown); Maasstad Hospital (Other)
Responsible Party: Principal Investigator, Pravesh S. Gadjradj, PhD-candidate, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRace 108226
Record Dates: First submitted 2018-03-17; First posted 2018-03-29 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Stenoses, Spinal
Keywords: laminectomy; laminotomy; lumbar canal stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Laminectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small size interarcuair decompression (Experimental): Patients will undergo small size interarcuair decompression
  Interventions: Procedure: small size interarcuair decompression
- Laminectomy (Active Comparator): Patients will undergo laminectomy
  Interventions: Procedure: Laminectomy

INTERVENTIONS:
Procedure: small size interarcuair decompression — A median lumbar incision is made and the paravertebral muscles are dissected subperiosteally and retracted unilaterally or bilaterally. Decompression will be applied via decompression of the ligamentum flavum. The lateral recess will be opened bilaterally and a medial facetectomy will be performed in order maintain stability of the segments. Posterior ligaments will be spared. The wound will be closed in layers with or without a suction drain. Patients will be operated with a loupe magnification or microscope depending on the surgeon's preference.
  Arms: Small size interarcuair decompression
Procedure: Laminectomy — A median lumbar incision is made over the spinous processes, the laminae of the affected level(s) are exposed subperiosteally, and the supraspinous ligament will be incised. The spinous process is removed. The supra and interspinous ligament of the affected level is removed by drill or Kerrison punches. The lamen is removed of the affect level, leaving the facet joint intact. The lateral recess will be opened bilaterally and medial facetectomy will be performed in order to maintain stability of the segments. When a single level stenosis is present (e.g. L4-L5) both laminae L4 and L5 will be removed. The wound will be closed in layers with or without a suction drain. Patients will be operated with loupe magnification or microscope depending surgeon's preference.
  Arms: Laminectomy

SUMMARY:
Rationale: Minimally invasive techniques have gained popularity to decompress lumbar spinal stenosis in the elderly. However, high quality evidence based on randomised controlled trials are not available.

Objective: To investigate whether small size interarcuair decompression is more effective than conventional laminectomy in patients with intermittent neurogenic claudication caused by lumbar spinal stenosis. Study design: Double-blinded multi-centre randomised controlled trial Study population: In total 236 patients are to be included. The inclusion criteria are: subjects > 40 years of age with at least 12 weeks of complaints of intermittent neurogenic claudication based on MRI confirmed of LSS, with sufficient knowledge of the Dutch language.

Intervention: Small size interarcuair decompression versus conventional laminectomy.

Main study parameters/endpoints: Primary outcome is the Modified Roland Morris Questionnaire. Secondary outcomes are leg pain, back pain and a 6 minute walk test amongst others.

Nature and extent of the burden and risks associated with participation: based on available literature , it is believed that the risks associated with small size interarcuair decompression are no greater than that associated with a laminectomy, although these will be examined.

DETAILED DESCRIPTION:
Intermittent neurogenic claudication (INC) caused by a lumbar spinal canal stenosis (LSS) is the most frequent reason for spinal surgery in the elderly. Multiple, less invasive surgical techniques are applied without sufficient evidence for benefits for patients or society.

The classic symptoms of INC are leg pain, which can be exacerbated with prolonged walking and standing and/or lumbar extension, and is associated with back pain. Severe stenosis is common in the elderly spine with 30.4% of the population having severe stenosis. However, only 17.5% have complaints of INC.

Conservative treatment, such as physical therapy or pain medication, may give some relief of symptoms. However, surgical treatment is considered to be the gold standard for patients with INC caused by LSS. The first technique ever described to widen the lumbar spinal canal is the wide bony decompression (laminectomy), which is still a widely used technique. However, since INC is often accompanied by back pain, and this to post-operative back pain, it is hypothesized that a wide decompression is a ground for potential instability. Hence, less invasive techniques, such as interarcuair decompression, were developed and implemented.

Recent studies claim that a limited bony decompression is the new 'golden standard' therapy for patients with INC. Limited bony decompression is believed to give less muscle damage and thus a faster postoperative recovery. Furthermore, wide bony decompression (such as a laminectomy) is believed to result in lumbar instability and iatrogenic scoliosis. Performing a procedure with potential more complications in a - generally - elderly population could at least be described as doubtful. The assumption is often made that after a wide decompression recurrence of the complaints must be scarce. However, a (cost-) effectiveness study, which evaluates the effectiveness of small bony decompression compared to a 'classical' extensive bony decompression, has not been performed yet. The opinions on this matter are diverse. A laminectomy involves the removal of more bone and structures at the back of the spine which may result in longer hospitalization and loss of productivity, but it could also lead to spinal instability on the long term. However, the risk of an insufficient decompression may be higher, potentially leading to more reoperations.

By the means of this double-blinded, multi-center randomized controlled trial the investigators will determine the (cost-) effectiveness of a limited bony decompression compared to a wide bony decompression in patients with INC.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 weeks of complaints of INC
* Magnetic resonance imaging showing LSS
* Age >40 years of age
* Sufficient knowledge of the Dutch language
* Signed informed consent

Exclusion Criteria:

* History of lumbar spine surgery
* >2 lumbar levels operation or needed discectomy
* Degenerative spondylolisthesis > grade 1 (on a scale of 1 to 4), scoliosis or disc herniation
* ASA-classification >3
* Serious psychopathology
* Pregnancy
* Active malignancy
* Plans to move abroad during study period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change on the Modified Roland-Morris Disability Questionnaire | baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  This is a 24-point Dutch questionnaire that is designed to assess the physical disability in patients, due to lower back pain.

SECONDARY OUTCOMES:
Change on the Numeric Rating Scale for leg pain | baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  The pain intensity in both legs (affected and non-affected) will be rated on a 11-point scale.
Change on the Numeric Rating Scale for back pain | baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  The pain intensity in the back will be rated on a 11-point scale.
Changes on the timed-up and go test | baseline, 6 months, 12 months, 24 months and 48 months after surgery
  This time will be measured in seconds
Changes on the 6-minute walk test | baseline, 6 months, 12 months, 24 months and 48 months after surgery
  The endurance and distance will be measured.
Changes on Neurological examination | baseline, 6 months, 12 months, 24 months and 48 months after surgery
  Motor changes of lower muscles will be measured.
Changes on the Timed Chair-Stand-Test (TCST) | baseline, 6 months, 12 months, 24 months and 48 months after surgery
  The time between standing and sitting on a chair will be measured.
Changes on the Oswestry Disability Index | baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  The ODI is one of the principal condition-specific outcome measures used in the management of spinal disorders.
Changes on Functional lumbar x-rays | baseline, 6 weeks
  A functional X-ray will be obtained from all patients X-ray will be made from AP and lateral position to assess spondylolisthesis. Degenerative spondylilolisthesis is defined as a vertebral slip of at least 3 mm.
Perceived recovery | 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  o measure the perceived recovery a seven-point Likert scale will be used. The score on this scale vary from 'completely recovered' to 'worse than ever'.
Patient satisfaction | 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  To measure patient satisfaction a seven-point Likert scale will be used. The score on this scale vary from 'completely satisfied with current symptoms' to 'completely dissatisfied with current symptoms'.
Changes on the SF-36 | Baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  The SF-36 will be used as a generic quality-of-life questionnaire. The SF-36 questionnaire has been validated and found reliable for low back pain.
Complications | 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  A systematic assessment of complications (including wound infection, deep venous thrombosis, urine tract infection, hematoma, and progressive neurological deficit) will be recorded out by the surgeon and research nurse, and these data are to be extracted from the patient chart. Moreover, surgeons will be asked for perioperative complications
Changes on the EuroQoL (EQ-5D) | Baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  The EuroQoL (EQ-5D) will be used for the cost utility analysis. The tool measures five dimensions: mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each dimension consists of one item, while five levels are distinguished (no, slight, moderate, severe problems, unable to do)
Costs of treatment measured using cost questionnaires filled out by the patients | Baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months and 48 months after surgery
  Cost questionnaires will be completed at the prescribed measurements. Hospitalisation for surgery will be registered using the case record forms. Other health care utilization (including physiotherapy, visits to GP and specialists, nursing care and medication), patient costs, and absenteeism from work will be measured using cost questionnaires filled out by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Biswadjiet Harhangi, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
After final publication of manuscript the data set will be available from the authors or journal of publication. Anonymized clinical data will be available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After final publication of manuscript without time limit.
Access Criteria: Anonymized

REFERENCES:
- [Derived] Arjun Sharma J, Gadjradj PS, Peul WC, van Tulder MW, Moojen WA, Harhangi BS; SIZE-study group. SIZE study: study protocol of a multicentre, randomised controlled trial to compare the effectiveness of an interarcuair decompression versus extended decompression in patients with intermittent neurogenic claudication caused by lumbar spinal stenosis. BMJ Open. 2020 Oct 6;10(10):e036818. doi: 10.1136/bmjopen-2020-036818. PMID 33028548